CLINICAL TRIAL: NCT03062280
Title: A Phase III Extension Study of Efficacy, Safety and Tolerability of Chronocort® in the Treatment of Congenital Adrenal Hyperplasia
Brief Title: A Study of the Efficacy, Safety and Tolerability of Chronocort in Treating CAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-006
Record Dates: First submitted 2016-08-22; First posted 2017-02-23 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Extension study
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chronocort® (Experimental): Chronocort® modified release hydrocortisone
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Modified release hydrocortisone

SUMMARY:
Subjects completing study DIUR-005 and those who have already completed study DIUR-003 will be offered the opportunity either to continue Chronocort® therapy or to switch from their current glucocorticoid therapy to Chronocort® in this open-label study.

DETAILED DESCRIPTION:
All subjects will have a screening visit prior to the baseline assessment to allow DIUR-006 procedures to be fully explained and informed consent to be given by the subject. For subjects from DIUR-003 this screening visit will include safety blood tests. Any subjects not meeting the inclusion/exclusion criteria following these blood tests will be not be entered into the study.

All subjects will then return for the baseline visit. For subjects entering from study DIUR-003 the full set of baseline assessments will be completed, including 2 blood samples (one at 09:00 and one at 13:00 hours) for 17-OHP and A4. For subjects entering from DIUR-005, test results from their last visit in the feeder study (Visit 4) will be used for this baseline assessment, with the 09:00 and 13:00 hour results taken from the 24-hour hormone profiles conducted at the visit. Any subjects not meeting the inclusion/exclusion criteria following these blood tests will be withdrawn from this study.

Once the baseline assessments are completed, the subjects will be given sufficient Chronocort® to use until the next visit at Week 4. Subjects from study DIUR-005 who were previously on Chronocort® will continue on the same dose of Chronocort® that they were receiving at the end of the feeder study. Subjects from study DIUR-005 on standard therapy and subjects from study DIUR-003 will have their initial dose of Chronocort® determined using the hydrocortisone equivalent of baseline therapy.

All subjects will return to the study centre at 4, 12 and 24 weeks after starting study DIUR-006 for additional blood tests and dose titration, if necessary. Visits thereafter will take place at 6-monthly intervals. If there is a change of dose, an interim visit or phone call will be needed inbetween the 6-monthly visits.

All subjects will receive telephone calls at 3 monthly intervals, and unscheduled visits will be arranged if necessary. Subjects will also be provided with Chronocort® supplies from the study pharmacy at 3-monthly or 6-monthly intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with CAH who have successfully completed a clinical trial with the current formulation of Chronocort®.
2. Provision of signed written informed consent.

Exclusion Criteria:

1. Co-morbid condition requiring daily administration of a medication (or use of any medications/supplements) that interferes with the metabolism of glucocorticoids.
2. Clinical or biochemical evidence of hepatic or renal disease. Creatinine over twice the ULN or elevated liver function tests (ALT or AST >2 times ULN]).
3. Females who are pregnant or lactating.
4. Subjects on regular daily inhaled, topical, nasal or oral steroids for any indication other than CAH.
5. History of malignancy (other than basal cell carcinoma successfully treated >6 months prior to entry into the study).
6. Subjects with a history of bilateral adrenalectomy.
7. Participation in another clinical trial of an investigational or licensed drug or device within the 3 months prior to inclusion in this study, except for another clinical trial with the current formulation of Chronocort®.
8. Subjects unable to comply with the requirements of the protocol.
9. Subjects who routinely work night shifts and so do not sleep during the usual nighttime hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Neurocrine UK Limited
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merke DP, Mallappa A, Arlt W, Brac de la Perriere A, Linden Hirschberg A, Juul A, Newell-Price J, Perry CG, Prete A, Rees DA, Reisch N, Stikkelbroeck N, Touraine P, Maltby K, Treasure FP, Porter J, Ross RJ. Modified-Release Hydrocortisone in Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2063-e2077. doi: 10.1210/clinem/dgab051. PMID 33527139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, open-label extension study. Participants who completed studies DIUR-003 (NCT01735617) or DIUR-005 (NCT02716818) were offered the opportunity to continue Chronocort® therapy in this study. After screening, all participants underwent a full set of baseline assessments before starting treatment in this extension study.
Groups:
- Chronocort®: Participants who entered immediately from Study DIUR-005 who were previously on Chronocort (modified release hydrocortisone) continued on the same dose of Chronocort that they had been receiving at the end of the feeder study. All other participants had their initial dose of Chronocort determined using the hydrocortisone equivalent of their current treatment (immediately prior to the baseline visit). Dosing was adjusted on an individual participant basis by investigators using symptoms and signs of disease with 17-hydroxyprogesterone (17-OHP) and androstenedione evaluation to guide dose adjustment.
Period: Overall Study
Arm/Group | Chronocort®
Started | 91
Completed | 69 (Completing the study is defined as being on-study when the study closed.)
Not Completed | 22
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Fertility Treatment | 2
Not completed — Physician Decision | 2
Not completed — Pregnancy | 5
Not completed — Withdrawal by Subject | 11

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort.
Groups:
- Chronocort®: Participants who entered immediately from Study DIUR-005 who were previously on Chronocort (modified release hydrocortisone) continued on the same dose of Chronocort that they had been receiving at the end of the feeder study. All other participants had their initial dose of Chronocort determined using the hydrocortisone equivalent of their current treatment (immediately prior to the baseline visit). Dosing was adjusted on an individual participant basis by investigators using symptoms and signs of disease with 17-OHP and androstenedione evaluation to guide dose adjustment.
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (11.76)
Age, Customized [Count of Participants; unit: Participants]
  >=18-<30 Years | 30
  >=30-<50 Years | 44
  >=50-<70 Years | 17
  >=70 Years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 89
  Asian | 0
  Black or African American | 0
  American Indian or Alaska native | 0
  Other | 2
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 162 (9.87)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 75.58 (16.091)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/square meter (m^2)] | 28.802 (5.6692)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.798 (0.2099)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 91.54 (14.810)
Time Since Congenital Adrenal Hyperplasia (CAH) Diagnosis [Mean (Standard Deviation); unit: years] | 35.76 (11.565)
Number of Participants Hospitalized Within the Last 12 Months Prior to Enrolment [Count of Participants; unit: Participants]
  Yes | 6
  No | 85
Number of Participants With Adrenal Crises in the Last Year [Count of Participants; unit: Participants]
  None | 86
  One | 5
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 70.6 (10.79)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 120.4 (13.92)
Pulse Rate [Mean (Standard Deviation); unit: beats/minute] | 71.1 (12.16)
Respiratory Rate [Mean (Standard Deviation); unit: breaths/minute] | 16.3 (2.85)
Body Temperature [Mean (Standard Deviation); unit: degrees Celsius (°C)] | 36.44 (0.427)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability - Number of Participants With Adrenal Insufficiency
Description: Safety and tolerability of Chronocort® over time, as assessed by signs and symptoms of adrenal insufficiency or over-treatment throughout the study. Signs and symptoms of adrenal insufficiency included sudden weight loss, sudden weight gain, lack of appetite, increased appetite, nausea, vomiting, headache, blurred vision, fatigue, weakness, dizziness, light-headedness, syncope, sleeping difficulties and increased acne. Number of participants who experienced adrenal insufficiency due to glucocorticoid (GC) over replacement and under replacement are reported.
Time Frame: Up to approximately 5 years and 11 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Participants
  Due to GC over-replacement | 25
  Due to GC under-replacement | 41

2. Primary Outcome: Safety and Tolerability - Number of Participants Who Used Sick Day Medication
Description: Safety and tolerability of Chronocort, as assessed by number of participants who used sick day medication throughout the study. Data are presented for number of participants taking medication from sick day packs and number of participants taking medication that was not from sick day packs.
Time Frame: Up to approximately 5 years and 11 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Participants
  Participants Taking Medication From Sick Day Packs | 79
  Participants Taking Medication That Was Not From Sick Day Packs | 47

3. Primary Outcome: Safety and Tolerability - Number of Participants Who Experienced at Least One Adrenal Crisis
Description: Safety and tolerability of Chronocort, as assessed by the number of participants who experienced adrenal crises throughout the study. Adrenal crisis was defined as follows: a) Major impairment of general health with at least two of the following signs/symptoms: Hypotension (systolic blood pressure <100 mmHg); Nausea or vomiting; Severe fatigue; Fever; Somnolence; Hyponatraemia (<132 mmol/L) or hyperkalaemia (as judged by characteristic electrocardiogram [ECG] changes); Hypoglycaemia and b) Parenteral glucocorticoid (hydrocortisone) administration followed by clinical improvement: Grade 1: outpatient care only; Grade 2: hospital care (general ward); Grade 3: admission to intensive care unit; Grade 4: death from adrenal crisis (with or without parenteral glucocorticoid administration).
Time Frame: Up to approximately 5 years and 11 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Participants | 7

4. Primary Outcome: Safety and Tolerability - Number of Participants With Adverse Events (AEs)
Description: Safety and tolerability of Chronocort, as assessed by the number of participants with at least 1 AE per specified AE category throughout the study. An AE was any untoward medical occurrence in a participant administered the study drug that did not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, was a congenital anomaly or birth defect, was infection that required treatment parenteral antibiotics, other important medical events which based on medical or scientific judgement might jeopardize the participants, or might require medical or surgical intervention to prevent any of the above. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to approximately 5 years and 11 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Participants
  Any AE | 90
  Any AE causally related to Chronocort | 37
  Any AE leading to sick day rules | 80
  Any AE leading to sick day rules causally related to Chronocort | 1
  Any AE leading to adrenal crisis | 7
  Any AE leading to adrenal crisis causally related to Chronocort | 0
  Any AE of unexpected therapeutic benefit | 21
  Any AE of unexpected therapeutic benefit causally related to Chronocort | 20
  Any AE leading to death | 1
  Any AE leading to death causally related to Chronocort | 0
  Any AE leading to discontinuation | 6
  Any AE leading to discontinuation causally related to Chronocort | 3
  Any serious adverse event (SAE) | 28
  Any SAE causally related to Chronocort | 2
  Any SAE leading to discontinuation | 0
  Any severe AE | 24
  Any severe AE causally related to Chronocort | 0
  Any AE associated with a dose increase | 6
  Any AE associated with a dose increase causally related to Chronocort | 2
  Any AE associated with a dose decrease | 7
  Any AE associated with a dose decrease causally related to Chronocort | 5
  Any AE associated with a dose interruption | 9
  Any AE associated with a dose interruption causally related to Chronocort | 0

5. Primary Outcome: Safety Laboratory Assessments - Number of Participants With a Shift in Laboratory Parameters Baseline Values to the Maximum Values
Description: Safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline in safety laboratory assessments throughout the study. Participants with a parameter value that shifted from baseline (within reference range) to a value above the reference range for a maximum value on-treatment.
Time Frame: Baseline up to approximately 5 years and 11 months
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. Number analyzed for each parameter = participants with a normal parameter value (within reference range) at baseline and also with at least one on-treatment value.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 87
Participants
  Red Blood Cell Count: number analyzed (Participants) | 77
  Red Blood Cell Count: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 6
  Red Blood Cell Count: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 71
  Haemoglobin: number analyzed (Participants) | 71
  Haemoglobin: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 5
  Haemoglobin: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 66
  Haematocrit: number analyzed (Participants) | 75
  Haematocrit: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 5
  Haematocrit: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 70
  Red cell distribution width: number analyzed (Participants) | 70
  Red cell distribution width: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 17
  Red cell distribution width: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 53
  Mean corpuscular volume: number analyzed (Participants) | 85
  Mean corpuscular volume: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 3
  Mean corpuscular volume: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 82
  Mean cell haemoglobin: number analyzed (Participants) | 82
  Mean cell haemoglobin: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 6
  Mean cell haemoglobin: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 76
  Mean cell haemoglobin concentration: number analyzed (Participants) | 82
  Mean cell haemoglobin concentration: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Mean cell haemoglobin concentration: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 81
  Platelet count: number analyzed (Participants) | 81
  Platelet count: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 3
  Platelet count: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 78
  Total White Blood Cell Count: number analyzed (Participants) | 82
  Total White Blood Cell Count: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 10
  Total White Blood Cell Count: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 72
  Lymphocyte count absolute: number analyzed (Participants) | 79
  Lymphocyte count absolute: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Lymphocyte count absolute: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 78
  Lymphocyte count percentage (%): number analyzed (Participants) | 64
  Lymphocyte count percentage (%): Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 9
  Lymphocyte count percentage (%): No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 55
  Monocyte count absolute: number analyzed (Participants) | 78
  Monocyte count absolute: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 0
  Monocyte count absolute: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 78
  Monocyte count %: number analyzed (Participants) | 83
  Monocyte count %: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 4
  Monocyte count %: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 79
  Neutrophil count absolute: number analyzed (Participants) | 78
  Neutrophil count absolute: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 8
  Neutrophil count absolute: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 70
  Neutrophil count %: number analyzed (Participants) | 72
  Neutrophil count %: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 15
  Neutrophil count %: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 57
  Basophil count absolute: number analyzed (Participants) | 83
  Basophil count absolute: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 0
  Basophil count absolute: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 83
  Basophil count %: number analyzed (Participants) | 82
  Basophil count %: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 0
  Basophil count %: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 82
  Eosinophil count absolute: number analyzed (Participants) | 76
  Eosinophil count absolute: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 7
  Eosinophil count absolute: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 69
  Eosinophil count %: number analyzed (Participants) | 81
  Eosinophil count %: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 12
  Eosinophil count %: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 69
  Sodium: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Sodium: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 86
  Potassium: number analyzed (Participants) | 85
  Potassium: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 0
  Potassium: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 85
  Chloride: number analyzed (Participants) | 76
  Chloride: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 7
  Chloride: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 69
  Total carbon dioxide: number analyzed (Participants) | 80
  Total carbon dioxide: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Total carbon dioxide: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 79
  Total calcium: number analyzed (Participants) | 84
  Total calcium: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Total calcium: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 83
  Total magnesium: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 2
  Total magnesium: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 85
  Inorganic phosphorus: number analyzed (Participants) | 70
  Inorganic phosphorus: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 5
  Inorganic phosphorus: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 65
  Creatinine: number analyzed (Participants) | 77
  Creatinine: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 2
  Creatinine: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 75
  Blood urea nitrogen: number analyzed (Participants) | 85
  Blood urea nitrogen: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Blood urea nitrogen: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 84
  Fasting glucose: number analyzed (Participants) | 72
  Fasting glucose: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 23
  Fasting glucose: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 49
  Uric acid: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 2
  Uric acid: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 85
  Total protein: number analyzed (Participants) | 61
  Total protein: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Total protein: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 60
  Albumin: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 2
  Albumin: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 85
  Alkaline phosphatase: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 2
  Alkaline phosphatase: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 85
  Alanine transaminase (ALT) / glutamate-pyruvate transaminase (GPT): Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 2
  Alanine transaminase (ALT) / glutamate-pyruvate transaminase (GPT): No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 85
  Aspartate aminotransferase (AST) / glutamic oxaloacetic transaminase (GOT): Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 3
  Aspartate aminotransferase (AST) / glutamic oxaloacetic transaminase (GOT): No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 84
  Total creatine kinase: number analyzed (Participants) | 85
  Total creatine kinase: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 14
  Total creatine kinase: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 71
  Lactate dehydrogenase: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 0
  Lactate dehydrogenase: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 87
  Total bilirubin: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 7
  Total bilirubin: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 80
  Direct bilirubin: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 1
  Direct bilirubin: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 86
  Total cholesterol: number analyzed (Participants) | 67
  Total cholesterol: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 36
  Total cholesterol: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 31
  High Density Lipoprotein (HDL) cholesterol: number analyzed (Participants) | 85
  High Density Lipoprotein (HDL) cholesterol: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 0
  High Density Lipoprotein (HDL) cholesterol: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 85
  Low density lipoprotein (LDL) cholesterol: number analyzed (Participants) | 34
  Low density lipoprotein (LDL) cholesterol: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 24
  Low density lipoprotein (LDL) cholesterol: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 10
  Triglycerides: number analyzed (Participants) | 84
  Triglycerides: Shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 12
  Triglycerides: No shift from pre-Chronocort baseline within reference range to above reference range on-treatment | 72

6. Primary Outcome: Safety Laboratory Assessments - Number of Participants With a Shift in Laboratory Parameters Baseline Values to the Minimum Values
Description: Safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline in safety laboratory assessments throughout the study. Participants with a parameter value that shifted from baseline (within reference range) to a value below the reference range for a minimum value on-treatment.
Time Frame: Baseline up to approximately 5 years and 11 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 87
Participants
  Red Blood Cell Count: number analyzed (Participants) | 77
  Red Blood Cell Count: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 5
  Red Blood Cell Count: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 72
  Haemoglobin: number analyzed (Participants) | 71
  Haemoglobin: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 13
  Haemoglobin: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 58
  Haematocrit: number analyzed (Participants) | 75
  Haematocrit: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 12
  Haematocrit: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 63
  Red cell distribution width: number analyzed (Participants) | 70
  Red cell distribution width: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 1
  Red cell distribution width: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 69
  Mean corpuscular volume: number analyzed (Participants) | 85
  Mean corpuscular volume: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 3
  Mean corpuscular volume: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 82
  Mean cell haemoglobin: number analyzed (Participants) | 82
  Mean cell haemoglobin: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 5
  Mean cell haemoglobin: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 77
  Mean cell haemoglobin concentration: number analyzed (Participants) | 82
  Mean cell haemoglobin concentration: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 13
  Mean cell haemoglobin concentration: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 69
  Platelet count: number analyzed (Participants) | 81
  Platelet count: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 1
  Platelet count: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 80
  Total White Blood Cell Count: number analyzed (Participants) | 82
  Total White Blood Cell Count: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 8
  Total White Blood Cell Count: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 74
  Lymphocyte count absolute: number analyzed (Participants) | 79
  Lymphocyte count absolute: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Lymphocyte count absolute: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 79
  Lymphocyte count %: number analyzed (Participants) | 64
  Lymphocyte count %: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 12
  Lymphocyte count %: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 52
  Monocyte count absolute: number analyzed (Participants) | 78
  Monocyte count absolute: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 10
  Monocyte count absolute: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 68
  Monocyte count %: number analyzed (Participants) | 83
  Monocyte count %: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Monocyte count %: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 83
  Neutrophil count absolute: number analyzed (Participants) | 78
  Neutrophil count absolute: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 10
  Neutrophil count absolute: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 68
  Neutrophil count %: number analyzed (Participants) | 72
  Neutrophil count %: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 10
  Neutrophil count %: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 62
  Basophil count absolute: number analyzed (Participants) | 83
  Basophil count absolute: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Basophil count absolute: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 83
  Basophil count %: number analyzed (Participants) | 82
  Basophil count %: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Basophil count %: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 82
  Eosinophil count absolute: number analyzed (Participants) | 76
  Eosinophil count absolute: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 13
  Eosinophil count absolute: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 63
  Eosinophil count %: number analyzed (Participants) | 81
  Eosinophil count %: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Eosinophil count %: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 81
  Sodium: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 6
  Sodium: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 81
  Potassium: number analyzed (Participants) | 85
  Potassium: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 4
  Potassium: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 81
  Chloride: number analyzed (Participants) | 76
  Chloride: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 1
  Chloride: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 75
  Total carbon dioxide: number analyzed (Participants) | 80
  Total carbon dioxide: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 3
  Total carbon dioxide: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 77
  Total calcium: number analyzed (Participants) | 84
  Total calcium: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 4
  Total calcium: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 80
  Total magnesium: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Total magnesium: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 87
  Inorganic phosphorus: number analyzed (Participants) | 70
  Inorganic phosphorus: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 7
  Inorganic phosphorus: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 63
  Creatinine: number analyzed (Participants) | 77
  Creatinine: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 12
  Creatinine: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 65
  Blood urea nitrogen: number analyzed (Participants) | 85
  Blood urea nitrogen: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 3
  Blood urea nitrogen: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 82
  Fasting glucose: number analyzed (Participants) | 72
  Fasting glucose: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 4
  Fasting glucose: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 68
  Uric acid: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 4
  Uric acid: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 83
  Total protein: number analyzed (Participants) | 61
  Total protein: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 4
  Total protein: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 57
  Albumin: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Albumin: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 87
  Alkaline phosphatase: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 2
  Alkaline phosphatase: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 85
  Alanine transaminase (ALT) / glutamate-pyruvate transaminase (GPT): Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Alanine transaminase (ALT) / glutamate-pyruvate transaminase (GPT): No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 87
  Aspartate aminotransferase (AST) / glutamic oxaloacetic transaminase (GOT): Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Aspartate aminotransferase (AST) / glutamic oxaloacetic transaminase (GOT): No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 87
  Total creatine kinase: number analyzed (Participants) | 85
  Total creatine kinase: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Total creatine kinase: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 85
  Lactate dehydrogenase: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Lactate dehydrogenase: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 87
  Total bilirubin: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Total bilirubin: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 87
  Direct bilirubin: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Direct bilirubin: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 87
  Total cholesterol: number analyzed (Participants) | 67
  Total cholesterol: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 3
  Total cholesterol: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 64
  High Density Lipoprotein (HDL) cholesterol: number analyzed (Participants) | 85
  High Density Lipoprotein (HDL) cholesterol: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 4
  High Density Lipoprotein (HDL) cholesterol: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 81
  Low density lipoprotein (LDL) cholesterol: number analyzed (Participants) | 34
  Low density lipoprotein (LDL) cholesterol: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 4
  Low density lipoprotein (LDL) cholesterol: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 30
  Triglycerides: number analyzed (Participants) | 84
  Triglycerides: Shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 0
  Triglycerides: No shift from pre-Chronocort baseline within reference range to below reference range on-treatment | 84

7. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - Diastolic Blood Pressure
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - Diastolic blood pressure.
Time Frame: Baseline, Month 30
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort. 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
mmHg | 2.7 (11.34)

8. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - Systolic Blood Pressure
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - Systolic blood pressure.
Time Frame: Baseline, Month 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
mmHg | -0.1 (12.81)

9. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - Pulse Rate
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - Pulse rate.
Time Frame: Baseline, Month 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
beats/minute | 0.2 (12.38)

10. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - Respiratory Rate
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - Respiratory rate.
Time Frame: Baseline, Month 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
breaths/minute | -0.2 (3.41)

11. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - Body Temperature
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - body temperature.
Time Frame: Baseline, Month 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
°C | 0.03 (0.464)

12. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - Body Weight
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - Body Weight.
Time Frame: Baseline, Month 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
kg | 0.14 (6.115)

13. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - BMI
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - BMI.
Time Frame: Baseline, Month 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
kg/m^2 | 0.086 (2.4248)

14. Primary Outcome: Safety and Tolerability - Change From Pre-Chronocort Baseline to Month 30 in Vital Signs - Waist Circumference
Description: Long-term safety and tolerability of Chronocort, as assessed by change from pre-Chronocort baseline to Month 30 in vital signs - Waist circumference.
Time Frame: Baseline, Month 30
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Chronocort®
Number analyzed (Participants) | 70
cm | 1.95 (7.1028)

15. Secondary Outcome: Total Daily Dose of Chronocort in Milligrams (mg)/Day of Hydrocortisone During the Time Interval Baseline to Week 4 and Month 18 to Month 24
Description: Total daily dose was summarized in mg/day of hydrocortisone where 1 mg of Chronocort equals 1 mg of hydrocortisone. Baseline was defined as the first visit of Study DIUR-006 for all participants.
Time Frame: Baseline to Week 4 and Month 18-24
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort. 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Median (Full Range); unit: mg/day
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
mg/day
  Baseline to Week 4 | 30.00 [10.00 to 55.00]
  Month 18 - Month 24: number analyzed (Participants) | 83
  Month 18 - Month 24 | 20.00 [6.80 to 55.00]

16. Secondary Outcome: Total Daily Dose of Chronocort in mg/Day/m^2 of Hydrocortisone by BSA During the Time Interval Baseline to Week 4 and Month 18 to Month 24
Description: Total daily dose of Chronocort per BSA was summarized in mg/day/m^2 of hydrocortisone where 1 mg of Chronocort equals 1 mg of hydrocortisone. The BSA (m^2) was calculated from baseline values using the Dubois formula [weight (kg)^0.425] x [Height (cm)^0.725)] x 0.007184. Baseline was defined as the first visit of Study DIUR-006 for all participants.
Time Frame: Baseline to Week 4 and Month 18-24
Population: as for outcome 15
Measure: Median (Full Range); unit: mg/day/m^2
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
mg/day/m^2
  Baseline to Week 4 | 15.764 [6.28 to 30.6]
  Month 18 - Month 24: number analyzed (Participants) | 83
  Month 18 - Month 24 | 11.766 [4.30 to 26.74]

17. Secondary Outcome: Number of Participants Achieving Disease Control at 09:00 Hours and 13:00 Hours for 17-hydroxyprogesterone (17-OHP)
Description: Long-term efficacy of Chronocort, as assessed by participants achieving disease control at 09:00 hours and 13:00 hours for 17-OHP. Data are presented for the number of participants considered responders and non-responders. A participant was considered a responder if their results were in the optimal range (defined as 1.2 to 36.4 nanomoles [nmol]/liter [L]) for 17-OHP.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort. 'Number analyzed' signifies participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Participants
  09:00 17-OHP : Baseline: number analyzed (Participants) | 90
  09:00 17-OHP : Baseline: Responder | 51
  09:00 17-OHP : Baseline: Non-responder | 39
  09:00 17-OHP : Week 24: number analyzed (Participants) | 87
  09:00 17-OHP : Week 24: Responder | 54
  09:00 17-OHP : Week 24: Non-responder | 33
  13:00 17-OHP : Baseline: Responder | 64
  13:00 17-OHP : Baseline: Non-responder | 27
  13:00 17-OHP : Week 24: number analyzed (Participants) | 87
  13:00 17-OHP : Week 24: Responder | 64
  13:00 17-OHP : Week 24: Non-responder | 23

18. Secondary Outcome: Number of Participants Achieving Disease Control at 09:00 Hours and 13.00 Hours for Androstenedione (A4)
Description: Long-term efficacy of Chronocort, as assessed by participants achieving disease control at 09:00 hours and 13:00 hours for A4. Data are presented for the number of participants considered responders and non-responders. A participant was considered a responder if their results were in the reference range (defined as 1.4 to 5.2 nmol/L in males and 1.0 to 7.0 nmol/L in females) for A4.
Time Frame: Baseline and Week 24
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Participants
  09:00 A4 : Baseline: number analyzed (Participants) | 90
  09:00 A4 : Baseline: Responder | 48
  09:00 A4 : Baseline: Non-responder | 42
  09:00 A4 : Week 24: number analyzed (Participants) | 87
  09:00 A4 : Week 24: Responder | 49
  09:00 A4 : Week 24: Non-responder | 38
  13:00 A4 : Baseline: Responder | 43
  13:00 A4 : Baseline: Non-responder | 48
  13:00 A4 : Week 24: number analyzed (Participants) | 87
  13:00 A4 : Week 24: Responder | 39
  13:00 A4 : Week 24: Non-responder | 48

19. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Bone Turnover Markers - Osteocalcin
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in bone turnover markers (osteocalcin).
Time Frame: Baseline, Month 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: micrograms (µg)/L
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
micrograms (µg)/L
  Osteocalcin, Baseline | 19.486 (7.8596)
  Osteocalcin, Change at Month 24: number analyzed (Participants) | 75
  Osteocalcin, Change at Month 24 | 3.535 (10.4837)

20. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Bone Turnover Markers - C-Terminal Cross-linked Telopeptide (CTX)
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in bone turnover markers - CTX.
Time Frame: Baseline, Month 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: nanograms (ng)/L
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
nanograms (ng)/L
  CTX, Baseline | 540.1 (251.84)
  CTX, Change at Month 24: number analyzed (Participants) | 74
  CTX, Change at Month 24 | -43.6 (228.53)

21. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Total Testosterone
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in total testosterone.
Time Frame: Baseline, Month 24
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort. Overall number of participants analyzed = number of male or female participants with evaluable data for the outcome measure. 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Chronocort® - Males: Males Chronocort® modified release hydrocortisone Hydrocortisone: Modified release hydrocortisone
- Chronocort® - Females: Females Chronocort® modified release hydrocortisone Hydrocortisone: Modified release hydrocortisone
Arm/Group | Chronocort® - Males | Chronocort® - Females
Number analyzed (Participants) | 29 | 62
nmol/L
  Total Testosterone, Baseline | 17.1490 (8.64256) | 0.9535 (1.38750)
  Total Testosterone, Change at Month 24: number analyzed (Participants) | 24 | 51
  Total Testosterone, Change at Month 24 | -1.5850 (6.51899) | -0.2892 (1.11890)

22. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Fasting Insulin
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in fasting insulin.
Time Frame: Baseline, Month 24
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort. 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: picomoles (pmol)/L
Arm/Group | Chronocort®
Number analyzed (Participants) | 90
picomoles (pmol)/L
  Fasting insulin, Baseline | 77.8 (35.61)
  Fasting insulin, Change at Month 24: number analyzed (Participants) | 73
  Fasting insulin, Change at Month 24 | -6.1 (36.41)

23. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Fasting Glucose
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in fasting glucose.
Time Frame: Baseline, Month 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: millimoles (mmol)/L
Arm/Group | Chronocort®
Number analyzed (Participants) | 90
millimoles (mmol)/L
  Fasting glucose, Baseline | 5.09 (0.434)
  Fasting glucose, Change at Month 24: number analyzed (Participants) | 74
  Fasting glucose, Change at Month 24 | -0.02 (0.534)

24. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Glycated Hemoglobin (HbA1c)
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in HbA1c.
Time Frame: Baseline, Month 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
percentage of HbA1c
  HbA1c, Baseline | 5.17 (0.312)
  HbA1c, Change at Month 24: number analyzed (Participants) | 75
  HbA1c, Change at Month 24 | 0.12 (0.235)

25. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in High Sensitivity C-reactive Protein (hsCRP)
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in hsCRP.
Time Frame: Baseline, Month 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
mg/L
  hsCRP, Baseline | 1.78 (5.010)
  hsCRP, Change at Month 24: number analyzed (Participants) | 75
  hsCRP, Change at Month 24 | 0.56 (6.290)

26. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Plasma Renin Activity (PRA)
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in PRA.
Time Frame: Baseline, Month 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/liter (L)/second
Arm/Group | Chronocort®
Number analyzed (Participants) | 90
ng/liter (L)/second
  PRA, Baseline | 0.878 (0.9587)
  PRA, Change at Month 24: number analyzed (Participants) | 85
  PRA, Change at Month 24 | 0.010 (1.2575)

27. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Body Composition - Total Lean Mass
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in body composition (Dual energy X-ray absorptiometry [DEXA]) - total lean mass
Time Frame: Baseline, Month 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Chronocort®
Number analyzed (Participants) | 71
kg
  Total lean mass, Baseline | 45.819 (9.3395)
  Total lean mass, Change at Month 24: number analyzed (Participants) | 55
  Total lean mass, Change at Month 24 | -0.563 (2.9490)

28. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Body Composition - Bone Mineral Density
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in body composition (DEXA) - bone mineral density.
Time Frame: Baseline, Month 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: grams (g)/square centimeter (cm^2)
Arm/Group | Chronocort®
Number analyzed (Participants) | 65
grams (g)/square centimeter (cm^2)
  Bone Mineral Density, Baseline | 1.0940 (0.09288)
  Bone Mineral Density, Change at Month 24: number analyzed (Participants) | 53
  Bone Mineral Density, Change at Month 24 | -0.0008 (0.03620)

29. Secondary Outcome: Change From Pre-Chronocort Baseline at Month 24 in Body Composition - Total Fat Mass
Description: Long-term efficacy of Chronocort, as assessed by change from pre-Chronocort baseline at Month 24 in body composition (DEXA) - total fat mass
Time Frame: Baseline, Month 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Chronocort®: Participants who entered immediately from Study DIUR-005 who were previously on Chronocort (modified release hydrocortisone) continued on the same dose of Chronocort that they had been receiving at the end of the feeder study. All other participants had their initial dose of Chronocort determined using the hydrocortisone equivalent of their current treatment (immediately prior to the baseline visit). Dosing was adjusted on an individual participant basis by investigators using symptoms and signs of disease with 17-OHP and androstenedione evaluation to guide dose adjustment.
  German subjects have been excluded from this analysis group as DEXA scans were not performed at German sites.
Arm/Group | Chronocort®
Number analyzed (Participants) | 71
kg
  Total fat mass, Baseline | 27.943 (11.5289)
  Total fat mass, Change at Month 24: number analyzed (Participants) | 55
  Total fat mass, Change at Month 24 | 0.811 (5.3320)

30. Secondary Outcome: Change From Pre-Chronocort Baseline in Quality of Life - Medical Outcome Short Form Health Survey Form 36 (SF-36) Score at Months 12 and 18
Description: The SF-36 questionnaire has 36 questions composing the scale that represent 8 domains: 1) physical functioning, role physical, 2) bodily pain, 3) general health, 4) vitality, 5) social functioning, 6) role, 7) emotional, and 8) mental health. The scores for the 8 domains were combined into two summary scores: the physical component summary (PCS) score and the mental component summary (MCS) score. Scores of the first four health items (1 - 4) were aggregated to derive the PCS ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition. Scores of last four items (5 - 8) were aggregated to derive the MCS ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition.
Time Frame: Baseline, Months 12 and 18
Population: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort. 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. 'Number analyzed' signifies participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronocort®
Number analyzed (Participants) | 84
units on a scale
  MCS, Change at Month 12 | 0.362 (12.3736)
  MCS, Change at Month 18: number analyzed (Participants) | 83
  MCS, Change at Month 18 | 0.257 (11.7003)
  PCS, Change at Month 12 | 0.496 (5.7091)
  PCS, Change at Month 18: number analyzed (Participants) | 83
  PCS, Change at Month 18 | 0.516 (6.8678)

31. Secondary Outcome: Change From Pre-Chronocort Baseline in Quality of Life - Multidimensional Assessment of Fatigue (MAF) Global Fatigue Index (GFI) Score at Months 12 and 18
Description: MAF is a 16-item scale that measures fatigue according to 4 dimensions; degree and severity, distress that it causes, timing of fatigue, and its impact of various activities of daily living. The GFI score was calculated using a standard method specific to the MAF questionnaire. This combines the responses to the questionnaire to give one score ranging from 1 (no fatigue) to 50 (severe fatigue), with a higher score indicating more severe fatigue, fatigue distress, or impact on activities of daily living. Decreases from baseline indicate improvement.
Time Frame: Baseline, Months 12 and 18
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronocort®
Number analyzed (Participants) | 85
units on a scale
  GFI, Change at Month 12 | -1.76 (11.939)
  GFI, Change at Month 18: number analyzed (Participants) | 83
  GFI, Change at Month 18 | -2.21 (12.847)

32. Secondary Outcome: Change From Pre-Chronocort Baseline in Quality of Life - Standardized Health Questionnaire 5-Dimension (EQ-5D) Index Score and Visual Analogue Scale (VAS) Score at Months 12 and 18
Description: The EQ-5D questionnaire consists of 2 parts, the EQ-5D descriptive system and the EQ VAS. The descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression each with 5 problem levels (1-none to 5-extreme). The results from the dimensions were combined using a standard method specially designed for the EQ-5D questionnaire to give a single index value (EuroQol Research Foundation) with scores ranging from 0 (no problems) to 1 (extreme problems). The EQ VAS is a visual scale in which the participant gives a single score between 0 (worst health state) and 100 (best health state).
Time Frame: Baseline, Months 12 and 18
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronocort®
Number analyzed (Participants) | 85
units on a scale
  EQ-5D-5L Index Score, Change at Month 12 | -0.022 (0.1766)
  EQ-5D-5L Index Score, Change at Month 18: number analyzed (Participants) | 83
  EQ-5D-5L Index Score, Change at Month 18 | -0.004 (0.1641)
  EQ VAS Score, Change at Month 12 | 1.529 (16.8612)
  EQ VAS Score, Change at Month 18: number analyzed (Participants) | 83
  EQ VAS Score, Change at Month 18 | 1.819 (15.7218)

33. Secondary Outcome: Number of Participants With Dose Titrations
Description: Long-term efficacy of Chronocort, as assessed by number of participants with dose titrations. Data are presented for number of participants with a dose increase, dose decrease, both a dose increase, and a dose decrease or no dose titration at specified timepoints.
Time Frame: Baseline to Week 4 and Month 18
Population: Full Analysis Set. 'Number analyzed' signifies participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Chronocort®
Number analyzed (Participants) | 91
Participants
  Baseline to Week 4: Dose increase | 0
  Baseline to Week 4: Dose decrease | 0
  Baseline to Week 4: Had both a dose increase and a dose decrease | 0
  Baseline to Week 4: No dose titration | 91
  Month 18: number analyzed (Participants) | 83
  Month 18: Dose increase | 2
  Month 18: Dose decrease | 17
  Month 18: Had both a dose increase and a dose decrease | 0
  Month 18: No dose titration | 64

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration up to approximately 5 years and 11 months
Description: The Full Analysis Set included all participants who entered the extension study and who subsequently received at least 1 dose of Chronocort.
Arm/Group | Chronocort®
All-Cause Mortality (participants affected / at risk) | 1/91
Serious Adverse Events (participants affected / at risk) | 28/91
Other Adverse Events (participants affected / at risk) | 90/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Chronocort® (N=91)
Appendicitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (4)
Influenza (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Malignant haemangiopericytoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 3 (9)
Anxiety (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Brachiocephalic vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 3 (4)
Melaena (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (2) — At risk population was based on maternal or paternal exposure.
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 1 (1) — At risk population was based on maternal or paternal exposure.
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Blood potassium decreased (Investigations) | 2 (2)
Red blood cell microcytes (Investigations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Chronocort® (N=91)
Acute sinusitis (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 2/62 (4) — This is a sex-specific AE, only female participants were at risk.
Balanitis candida (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 10 (23)
COVID-19 (Infections and infestations) | 17 (18)
Candida infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 4 (8)
Device related infection (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 4 (4)
Fungal infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 23 (27)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 6 (6)
Gingivitis (Infections and infestations) | 2 (2)
Helicobacter infection (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 30 (54)
Localised infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 8 (12)
Nasopharyngitis (Infections and infestations) | 34 (105)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 4 (4)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 7 (7)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 9 (16)
Staphylococcal infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 11 (16)
Urinary tract infection (Infections and infestations) | 12 (13)
Viral infection (Infections and infestations) | 3 (4)
Vulval abscess (Infections and infestations) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Vulvovaginal candidiasis (Infections and infestations) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Vulvovaginal mycotic infection (Infections and infestations) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Vulvovaginitis (Infections and infestations) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Adrenal rest tumour of the testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/29 (1) — This is a sex-specific AE, only male participants were at risk.
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (2)
Allergy to chemicals (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Thyroid mass (Endocrine disorders) | 1 (1)
Thyroiditis subacute (Endocrine disorders) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (5)
Increased appetite (Metabolism and nutrition disorders) | 4 (4)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1)
Anticipatory anxiety (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (11)
Bipolar I disorder (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 10 (11)
Insomnia (Psychiatric disorders) | 20 (23)
Libido decreased (Psychiatric disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (3)
Stress (Psychiatric disorders) | 9 (16)
Ageusia (Nervous system disorders) | 2 (2)
Anosmia (Nervous system disorders) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 10 (12)
Circadian rhythm sleep disorder (Nervous system disorders) | 1 (1)
Clumsiness (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 15 (25)
Headache (Nervous system disorders) | 37 (66)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 5 (21)
Paraesthesia (Nervous system disorders) | 9 (9)
Paresthesia (Nervous system disorders) | 1 (1)
Poor quality sleep (Nervous system disorders) | 2 (3)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (4)
Syncope (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Cataract (Eye disorders) | 1 (2)
Dry eye (Eye disorders) | 1 (1)
Episcleritis (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 2 (2)
Optic ischaemic neuropathy (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 4 (5)
Vitreous floaters (Eye disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (3)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3)
Rebound tachycardia (Cardiac disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (6)
Peripheral venous disease (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (8)
Abdominal pain upper (Gastrointestinal disorders) | 10 (15)
Anal pruritus (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 27 (63)
Diverticulum (Gastrointestinal disorders) | 3 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 20 (26)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Oral disorder (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Teeth brittle (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 31 (48)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (5)
Rash (Skin and subcutaneous tissue disorders) | 8 (9)
Skin laxity (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (22)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4)
Limb mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (15)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 (4)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Azoospermia (Reproductive system and breast disorders) | 1/29 (1) — This is a sex-specific AE, only male participants were at risk.
Breast pain (Reproductive system and breast disorders) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3/62 (5) — This is a sex-specific AE, only female participants were at risk.
Endometrial hyperplasia (Reproductive system and breast disorders) | 3/62 (3) — This is a sex-specific AE, only female participants were at risk.
Gynaecomastia (Reproductive system and breast disorders) | 1/29 (1) — This is a sex-specific AE, only male participants were at risk.
Menometrorrhagia (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Menopausal symptoms (Reproductive system and breast disorders) | 2/62 (2) — This is a sex-specific AE, only female participants were at risk.
Menorrhagia (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Menstruation irregular (Reproductive system and breast disorders) | 8/62 (10) — This is a sex-specific AE, only female participants were at risk.
Metrorrhagia (Reproductive system and breast disorders) | 3/62 (4) — This is a sex-specific AE, only female participants were at risk.
Ovarian cyst (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Testicular mass (Reproductive system and breast disorders) | 2/29 (2) — This is a sex-specific AE, only male participants were at risk.
Testicular pain (Reproductive system and breast disorders) | 1/29 (1) — This is a sex-specific AE, only male participants were at risk.
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/62 (2) — This is a sex-specific AE, only female participants were at risk.
Vulvar melanosis (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/62 (1) — This is a sex-specific AE, only female participants were at risk.
BRCA1 gene mutation (Congenital, familial and genetic disorders) | 1 (1)
Asthenia (General disorders) | 14 (21)
Chills (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 43 (106)
Feeling abnormal (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Injection site dermatitis (General disorders) | 1 (1)
Malaise (General disorders) | 11 (16)
Oedema mucosal (General disorders) | 1 (3)
Oedema peripheral (General disorders) | 5 (8)
Pain (General disorders) | 2 (2)
Performance status decreased (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 2 (2)
Pyrexia (General disorders) | 37 (66)
Swelling (General disorders) | 1 (1)
Swelling face (General disorders) | 2 (2)
Therapeutic response unexpected (General disorders) | 27 (46)
Vaccination site pain (General disorders) | 1 (1)
Vaccination site swelling (General disorders) | 1 (1)
Blood androstenedione increased (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3)
Blood glucose increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Blood testosterone decreased (Investigations) | 2 (2)
Blood testosterone increased (Investigations) | 3 (3)
Bone density decreased (Investigations) | 3 (3)
Bone density increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Eosinophil count decreased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 3 (3)
Haemoglobin decreased (Investigations) | 4 (4)
Heart rate decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Low density lipoprotein increased (Investigations) | 4 (5)
Occult blood (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 2 (2)
Red blood cell microcytes (Investigations) | 1 (1)
Renin decreased (Investigations) | 2 (2)
Renin increased (Investigations) | 4 (4)
Weight increased (Investigations) | 3 (3)
White blood cell count increased (Investigations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (3)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3)
Heat stroke (Injury, poisoning and procedural complications) | 2 (2)
Hypobarism (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 5/62 (6) — This is a sex-specific AE, only female participants were at risk.
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Paternal exposure before pregnancy (Injury, poisoning and procedural complications) | 3/29 (5) — This is a sex-specific AE, only male participants were at risk.
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2)
COVID-19 immunisation (Surgical and medical procedures) | 17 (24)
Gingival graft (Surgical and medical procedures) | 1 (2)
Tooth extraction (Surgical and medical procedures) | 3 (3)
Educational problem (Social circumstances) | 2 (2)
Family stress (Surgical and medical procedures) | 1 (1)
Impaired work ability (Social circumstances) | 1 (1)
Physical assault (Social circumstances) | 1 (1)
Stress at work (Social circumstances) | 2 (3)
Ear deformity acquired (Ear and labyrinth disorders) | 1 (2)
Foreign body sensation in eyes (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
c-reactive protein decreased (Investigations) | 1 (1)
Alcohol intolerance (Metabolism and nutrition disorders) | 1 (1)
Gluten sensitivity (Metabolism and nutrition disorders) | 1 (1)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1/29 (1) — This is a sex-specific AE, only male participants were at risk.
Blister (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor & PI will prepare of manuscripts. Comments on publications will be considered by authors. Publications will not include company confidential details without Sponsor permission. Summary data may be announced to comply with Financial & Regulatory Authorities, while ensuring this will not impact the investigator's ability to publish. Announcements made prior to publication will be reviewed & approved by PI. Data from individual sites will only be published under exceptional circumstances.

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03062280/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT03062280/SAP_001.pdf